CLINICAL TRIAL: NCT01403597
Title: Clinical Evaluation of the Impact of Non-ablative and Fractional Ablative Combination Treatment: a Prospective, Open Label, Single Group With Before-after Study Design
Brief Title: Evaluation of Non-ablative and Fractional Combination Treatment for Improvement in Skin's Appearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCP-1
Record Dates: First submitted 2011-07-20; First posted 2011-07-27 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Laser Therapy; Rejuvenation
Keywords: Skin wrinkling; Skin aging; Skin pigmentation
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): The defined areas for treatment are the entire face or at least two facial sub areas (e.g., peri-orbital and peri oral) with the combination of two devices where a total of 5 treatments every 4 weeks will be administered
  Interventions: Device: Refirme ST Applicator and Matrix RF Applicator

INTERVENTIONS:
Device: Refirme ST Applicator and Matrix RF Applicator — 5 treatments with combination of devices every 4 weeks to the facial (or sub facial regions).

SUMMARY:
The study is designed to determine the safety, efficacy, patient comfort and patient satisfaction of the combined treatment of Refirme ST and Matrix RF both devices approved under 510k clearances. The evaluations will include skin condition, physician/subject improvement assessment, and subject comfort and satisfaction score by questionnaires.

DETAILED DESCRIPTION:
The Refirme ST and the Matrix RF applicators are both FDA approved devices indicated for improvement of skin appearance. The Matrix RF applicator has FDA clearance for ablation, resurfacing of the skin, and for wrinkles treatment, whereas the Refirme-ST applicator has FDA clearance for non-invasive wrinkles treatment. The combined treatment of Refirme ST and Matrix RF is intended to improve skin appearance both by enhancement of collagen production as the result of the Refirme ST primary heating of the treated area and by causing ablation and resurfacing of the skin with the Matrix RF. In the current clinical setting, each applicator is used in a separate session although there is no contra-indication preventing the usage of these applicators in the same treatment session. A combined treatment in one session is believed to be more efficient and will be more time effective for the patient and therefore will have a commercial benefit for the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Have skin condition that requires ablation and resurfacing such as visible lines, pores, pigmentation, and elastosis that correlate to a score of 2 6 on the Fitzpatrick Classification of Wrinkling and Degree of Elastosis
* Age: At least 21 years of age and not older than 65 years of age
* Sex male or female
* For female candidates - post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide, or abstinence).
* Agrees to sign the Informed Consent
* Desire to improve their facial skin appearance
* Willingness to have photographs of the treated area taken that may be used for marketing and educational presentation and/or publications
* Willingness to follow the treatment and follow-up schedule and the post-treatment care
* Not planning to improve their skin appearance in a different procedure during the complete experimental period.

Exclusion Criteria:

* History of keloid scarring or of abnormal wound healing
* Suffering from current or history of significant skin conditions in the treated area or inflammatory skin conditions, including, but not limited to: excessive skin dryness, psoriasis, eczema, rash, rosacea (particularly severe open wound stage), indurate acne, varicella scars, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
* History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation
* Vascular lesion, tattoo or permanent make-up in the treated area
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breastfeeding.
* Suffering from hormonal imbalance, as per the Investigator's discretion.
* Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
* Having a permanent implant in the treated area, such as metal plates and screws, or an injected chemical substance.
* Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
* History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
* Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
* Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), or pertinent neurological disorders.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.
* Use of isotretinoin (Accutane®) within 6 months of treatment or during the study
* Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) one week before and after each treatment session
* Use of retinoids, antioxidants or skin nourishing supplements within 2 months of treatment or during the study.
* Having undergone any other surgery in the treated area within 6 months of treatment (or more if skin has not healed completely) or during the study
* Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion).
* Having received treatment with a light-based, radiofrequency or other devices within 3 month prior to treatment or during the study.
* Having received a facial dermabrasion or chemical peel treatment within 3 months of treatment or during the study.
* Having received Botox/collagen/fat injections or other methods of augmentation with injected or implanted material in the treated area within 3 months of treatment or during the study
* Having undergone a resurfacing procedure, face lift or eyelid surgery within a year of treatment or during the study
* Participation in a study of another device or drug within one month prior to enrollment or during the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety of treatment | 11 months
  The treatment will be considered safe if no cutaneous reactions (including excessive erythema and edema, blister formation, erosion, ulcer, scarring, infection, pruritis or allergic reactions) except of mild pigment can be detected at the site of treatment at the final follow up.
Efficacy of Treatment | 11 months
  The treatment will be considered efficacious if a result greater than ≥3 moderate to significant on GAI scale) of overall skin improvement will be marked at the final follow up

SECONDARY OUTCOMES:
Patient Satisfaction | 11 months
  The treatment will be considered satisfactory by the patient if a result ≥ 3 in the patient satisfaction scale will marked at the final follow up.
Patient Comfort | 11 months
  The treatment will be considered comfortable if a result ≥ 2 in the patient comfort assessment scale will marked at the end of at least 3/5 or 2/4 treatments.